CLINICAL TRIAL: NCT01898949
Title: BAT&DIT: Stimulation of Diet-Induced Thermogenesis by Cold-Exposure
Brief Title: Stimulation of Diet-Induced Thermogenesis by Cold-Exposure
Acronym: BAT&DIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Eric Ravussin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 10031
Record Dates: First submitted 2013-07-07; First posted 2013-07-15 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Thermogenesis; Brown Adipose Tissue
Keywords: Diet-induced thermogenesis; Cold-induced thermogenesis; Brown adipose tissue; Brown fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cold Exposure (Experimental)
  Interventions: Other: Cold Exposure

INTERVENTIONS:
Other: Cold Exposure — Participants will spend 20 minutes per day 5 times a week (workdays) in a cold room wearing light clothes (T-shirt, shorts and light shoes) for 4 weeks.

SUMMARY:
Human fat tissue is essentially white fat, the main function of which is to store excess energy intake, and to release it when necessary. Brown fat is far less abundant and is present in the body to burn fat (and thus energy) to generate heat to maintain body temperature around 96 degrees. This phenomenon is called thermogenesis. When humans are exposed to cold on a chronic basis, brown fat expands and becomes more active, and consequently burns more energy. The amount of brown fat is higher during winter, and daily short (20 minutes) exposures to cold might be sufficient to induce its activity.

We hypothesized that daily short term (20 minutes) exposure to a cold environment (4 °C) for four weeks increases adaptive BAT-mediated thermogenesis. CIT and DIT will be increased proportionally (the increase in CIT and DIT will be correlated).

DETAILED DESCRIPTION:
This study will have 3 phases:

Phase 1: baseline testing. This phase takes place at the beginning of the study to establish several physical, physiological and metabolic studies and includes measures of height, weight, body composition, sedentary and resting metabolic rate in a metabolic chamber as well as your metabolic and cardiac responses to cold.

Phase 2: cold exposure (treatment) phase. This phase is initiated immediately after phase 1 and will last 4 weeks. Each work day (Monday to Friday) subjects will have to spend 20 minutes in a cold room wearing light clothes.

Phase 3: post-treatment testing. The same physiological and metabolic studies measured at baseline will be repeated over 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Men between the ages of 18-35 years, inclusive
* Body mass index (BMI) between 18.5 and 25.0 kg/m2, inclusive, with a stable weight (<2kg variation) within the past 3-6 months
* Non smokers
* On no medication or recreational drugs
* Healthy as assessed by a standard self-reported screening health questionnaire
* Provide written informed consent

Exclusion Criteria:

* Smokers
* Individuals taking any medications
* Individuals taking any stimulants
* Individuals taking beta-blockers
* Individuals with diabetes or impaired fasting glucose as defined by theADA criteria, i.e. fasting plasma glucose concentration ≥ 5.6 mmol/L (100 mg/dl).
* Individuals with chronic alcohol consumption (> 3 drinks per day) or drug abuse
* Individuals unable to abstain from caffeinated beverage or alcohol the days of study
* Individuals with pacemakers or defibrillators
* Individuals with history of heart disease or history of stroke
* Individuals having a significant recent loss or gain of weight
* Individuals involved in regular (> 3 times per week), intense competitive sporting activities.
* Individuals involved in intensive exercise activity.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Energy Expenditure | After 4 weeks of cold exposure
  Change in energy expenditure is measured within 24 hours (acute) and after 4 weeks (chronic) of cold exposure with either bed-side calorimeter or whole-room calorimeter.

SECONDARY OUTCOMES:
Temperature | After 4 weeks of cold exposure
  Change in temperature acute (within 24 hours) and chronic (after 4 weeks) temperature from baseline as measured by either capsule (core body temperature) or infrared imaging (surface temperature).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ravussin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Lam YY, Redman LM, Smith SR, Bray GA, Greenway FL, Johannsen D, Ravussin E. Determinants of sedentary 24-h energy expenditure: equations for energy prescription and adjustment in a respiratory chamber. Am J Clin Nutr. 2014 Apr;99(4):834-42. doi: 10.3945/ajcn.113.079566. Epub 2014 Feb 5. PMID 24500151